CLINICAL TRIAL: NCT00072865
Title: A Phase II Study of Alimta and Carboplatin in the Treatment of Patients With Locally Advanced or Metastatic Breast Cancer
Brief Title: Pemetrexed and Carboplatin in Locally Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7771; H3E-MW-JMGJ
Record Dates: First submitted 2003-11-12; First posted 2003-11-13 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Breast Cancer; Neoplasm Metastasis
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Pemetrexed; Carboplatin

INTERVENTIONS:
Drug: Pemetrexed
Drug: Carboplatin

SUMMARY:
This is a nonrandomized study of pemetrexed plus carboplatin, with the primary objective of determining the efficacy of the combination in tumor reduction, in patients with locally advanced or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of locally advanced or metastatic breast cancer
* No prior chemotherapy for locally advanced or metastatic breast disease.
* Patient may have received prior adjuvant therapy finished greater than 1 year prior to enrollment.
* Adequate bone marrow, liver and kidney function
* RECIST criteria for disease status

Exclusion Criteria:

* Prior treatment with pemetrexed
* Pregnant or breast feeding
* Brain Metastasis
* unable or unwilling to take folic acid, vitamin B12 supplementation, or dexamethasone.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-06; Study Completion 2005-09

PRIMARY OUTCOMES:
antitumor activity

SECONDARY OUTCOMES:
duration of response;time to progressive disease;time to treatment failure

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Russia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Moscow, Russia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Saint Petersburg, Russia